CLINICAL TRIAL: NCT03011476
Title: Effect of Acetylcholinesterase Inhibitors on the Gait of the Patients With Parkinson Disease Characterized by Postural Instability and Gait Disturbance
Brief Title: Effect of Acetylcholinesterase Inhibitors on the Gait of the Patients With Parkinson Disease
Acronym: EASE-PIGD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyung Hee University Hospital (Other)
Responsible Party: Principal Investigator, Tae-Beom Ahn, Professor, Kyung Hee University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-08-030-003
Record Dates: First submitted 2016-12-27; First posted 2017-01-05 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donepezil (Active Comparator): dosage: 5mg, 10mg frequency: once a day duration: 12 weeks
  Interventions: Drug: Donepezil
- Placebos (Placebo Comparator): dosage: 5mg, 10mg frequency: once a day duration: 12 weeks
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Donepezil — 1. Start with 5 mg/day for 4 weeks
  2. Increased to 10 mg/day for 8 weeks
  Other Names: Aridone
  Arms: Donepezil
Drug: Placebos — 1. Start with 5 mg/day for 4 weeks
  2. Increased to 10 mg/day for 8 weeks
  Arms: Placebos

SUMMARY:
Cholinergic deficiency in the brain can be related to gait and balance problems in Parkinson disease (PD). Recent clinical trials suggested a beneficial role of acetylcholinesterase inhibitors (AchEI) on gait in PD. In this study, the investigators are planning to study the influence of AchEI on a brain network for gait and balance in PD. As gait problem is prominent in postural instability and gait disturbance (PIGD) subtype, this study will focus on the patients with PIGD phenotype.

DETAILED DESCRIPTION:
PD patients with PIGD subtype will be included.

1. Assessment:

   * Overall features of PD are assessed by Unified Parkinson Disease Rating Scale (UPDRS). Non-motor features including cognition will be assessed by standard scales. Gait and balance will be assessed by gait analysis system, which measures physiological parameters of gait such as velocity, variability and center of pressure. Positron emission tomography using 18F-fluorodeoxyglucose (FDG PET) will be done to brain activities related to gait and balance.
   * Clinical evaluation will be done at the baseline, 4th, 8th and 12th week
   * Gait analysis and FDG PET will be done at the baseline and 12th week
2. Drug dosage

   * For the first 4 weeks, 5 mg/day
   * Then, 10 mg/day for 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease diagnosed by United Kingdom Parkinson's disease Society Brain Bank Criteria
* Postural instability and gait disturbance phenotype
* Hoehn and Yahr stage ≤ 3
* Mini-Mental status examination ≥ 24

Exclusion Criteria:

* Significant motor complication affecting daily activities
* Drugs related to acetylcholine metabolism

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Positron emission tomography using 18F-flurodeoxyglucose | Metabolic change from Baseline at 12 weeks

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | Baseline assessment/ Follow-up assessment at 12th week
Unified Parkinson disease rating scale (UPDRS) | Baseline assessment/ Follow-up assessment at 4th, 8th and 12th week
Time-Up and Go | Baseline assessment/ Follow-up assessment at 4th, 8th and 12th week
Gait analysis | Baseline assessment/ Follow-up assessment at 4th, 8th and 12th week
  Composite measures of gait and balance

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Beom Ahn, MD, PhD, Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyung Hee Universtiy Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Henderson EJ, Lord SR, Brodie MA, Gaunt DM, Lawrence AD, Close JC, Whone AL, Ben-Shlomo Y. Rivastigmine for gait stability in patients with Parkinson's disease (ReSPonD): a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Neurol. 2016 Mar;15(3):249-58. doi: 10.1016/S1474-4422(15)00389-0. Epub 2016 Jan 13. PMID 26795874
- [Result] Henderson EJ, Lord SR, Close JC, Lawrence AD, Whone A, Ben-Shlomo Y. The ReSPonD trial--rivastigmine to stabilise gait in Parkinson's disease a phase II, randomised, double blind, placebo controlled trial to evaluate the effect of rivastigmine on gait in patients with Parkinson's disease who have fallen. BMC Neurol. 2013 Dec 3;13:188. doi: 10.1186/1471-2377-13-188. PMID 24299497
- [Result] Bohnen NI, Frey KA, Studenski S, Kotagal V, Koeppe RA, Scott PJ, Albin RL, Muller ML. Gait speed in Parkinson disease correlates with cholinergic degeneration. Neurology. 2013 Oct 29;81(18):1611-6. doi: 10.1212/WNL.0b013e3182a9f558. Epub 2013 Sep 27. PMID 24078735
- [Result] Bohnen NI, Muller ML, Koeppe RA, Studenski SA, Kilbourn MA, Frey KA, Albin RL. History of falls in Parkinson disease is associated with reduced cholinergic activity. Neurology. 2009 Nov 17;73(20):1670-6. doi: 10.1212/WNL.0b013e3181c1ded6. PMID 19917989
- [Result] Montero-Odasso M, Muir-Hunter SW, Oteng-Amoako A, Gopaul K, Islam A, Borrie M, Wells J, Speechley M. Donepezil improves gait performance in older adults with mild Alzheimer's disease: a phase II clinical trial. J Alzheimers Dis. 2015;43(1):193-9. doi: 10.3233/JAD-140759. PMID 25079803
- [Result] Stebbins GT, Goetz CG, Burn DJ, Jankovic J, Khoo TK, Tilley BC. How to identify tremor dominant and postural instability/gait difficulty groups with the movement disorder society unified Parkinson's disease rating scale: comparison with the unified Parkinson's disease rating scale. Mov Disord. 2013 May;28(5):668-70. doi: 10.1002/mds.25383. Epub 2013 Feb 13. PMID 23408503